CLINICAL TRIAL: NCT03229941
Title: CSP #599 - Transfusion Trigger After Operations in High Cardiac Risk Patients (TOP)
Brief Title: Transfusion Trigger After Operations in High Cardiac Risk Patients
Acronym: TOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 599
Record Dates: First submitted 2017-07-07; First posted 2017-07-26 (Actual); Results first posted 2025-09-05 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Myocardial Infarction; Coronary Revascularization; Acute Renal Failure
MeSH Terms: conditions — Myocardial Infarction; Acute Kidney Injury | interventions — Blood Transfusion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Restrictive (Experimental): Transfusion trigger: Hb<7gm/dl
  Interventions: Procedure: Blood Transfusion
- Liberal (Experimental): Transfusion trigger: Hb<10gm/dl
  Interventions: Procedure: Blood Transfusion

INTERVENTIONS:
Procedure: Blood Transfusion — Blood Transfusion

SUMMARY:
The goal of the proposed study is to determine whether a liberal transfusion strategy (transfusion trigger at Hb < 10 gm/dl) in Veterans at high cardiac risk who undergo major open vascular and general surgery operations is associated with decreased risk of adverse postoperative outcomes compared to a restrictive transfusion strategy (transfusion trigger at Hb < 7 gm/dl).

DETAILED DESCRIPTION:
Background: Despite the need for clinically appropriate use of blood products in the postoperative setting, blood transfusion practices are empiric and variable. In the absence of a physiologic test that can effectively guide transfusion-related decisions after an operative intervention, hemoglobin-based transfusion triggers have been suggested as clinical tools. Traditionally, clinicians have transfused patients to maintain hemoglobin (Hb) above a minimum (typically 10 gm/dl) level, in order to prevent adverse cardiac events and death. Recent randomized trials, however, have shown that restrictive transfusion policies (transfusion when Hb falls below 8 gm/dl or even lower) are well tolerated by specific patient populations. Furthermore, these trials have demonstrated that in some patient subsets reduced transfusion is associated with reduction in postoperative complications and death. Thus, guidelines have been developed emphasizing the need for a restrictive transfusion strategy in most stable hospitalized patients.

Despite the emerging enthusiasm with respect to the safety of restrictive transfusion strategies, high quality evidence on the value of such an approach in patients at high risk for postoperative adverse cardiac events remains scarce. This is a serious limitation of the current literature, as ischemic heart disease (IHD) is highly prevalent and represents the leading cause of mortality in this country, accounting for the death of one American every minute. Furthermore, there is evidence from small trials and secondary analyses that in this subset of patients withholding transfusion when Hb falls below 10 gm/dl increases the risk of death or myocardial infarction, suggesting that widespread use of restrictive transfusion policies may actually result in patient harm. This uncertainty on transfusion thresholds in high cardiac risk patients has created a knowledge gap that requires urgent attention. IHD is highly prevalent in patients with peripheral arterial disease (PAD), and myocardial infarction represents the leading cause of postoperative mortality in patients undergoing PAD-related surgical interventions. Furthermore, a substantial proportion of patients undergoing Vascular and General Surgery operations have history of prior IHD, making this patient population an ideal high cardiac risk group in which to analyze the effect of transfusion strategies. In order to address the knowledge gap of postoperative transfusion thresholds in patients at high risk for postoperative adverse cardiac events, the investigators propose the current study under the hypothesis that transfusion strategy will affect important postoperative outcomes after major surgical interventions in high cardiac risk patients.

Objectives: The goal of the proposed study is to determine whether a liberal postoperative transfusion strategy (transfusion trigger at Hb<10gm/dl) in patients at high risk for postoperative adverse cardiac events will reduce the risk of adverse postoperative outcomes after major vascular and general surgery operative interventions. The primary end point is the composite rate of all-cause mortality, acute myocardial infarction (MI), coronary revascularization, stroke, or acute renal failure within 90 days from the time of randomization. The secondary end points are rates of postoperative infectious complications (wound infections, pneumonia, and sepsis), and postoperative cardiac complications (new cardiac arrhythmias, congestive heart failure exacerbation, and cardiac arrest) at 90 days post-randomization; the composite rate of all-cause mortality, MI, coronary revascularization, stroke, or acute renal failure, within 30 days from the time of randomization; the length of hospital stay; and all-cause mortality up to one year after randomization.

Design: CSP #599 - TOP study is a randomized, intent-to-treat, two-arm, parallel design, single blind, multicenter trial. Vascular and General Surgery programs at Veterans Affairs Medical Centers with expertise in performing the operations of interest will be invited to participate and participants will be screened for enrollment using established inclusion/exclusion criteria. Enrolled participants will be randomized to one of the two arms; liberal (transfusion trigger at Hb < 10gm/dl) or restrictive (transfusion trigger at Hb < 7gm/dl). Consent for the study will be obtained prior to the index surgical intervention. Randomization will be performed postoperatively after the patient has a confirmed Hb < 10gm/dl. Assessments will be collected pre/post-operatively and at discharge, or at 30 days after randomization if the patient is still hospitalized. Follow up forms will be filled out during a clinic visit after the 30th and 90th post-randomization day. Patients who cannot present to the clinic will have a phone call for follow up. One year post-randomization mortality will be ascertained using electronic medical records, phone follow-up, and search of the national death index.

Sample Size and Study Duration: This study will randomize 1520 participants undergoing major vascular and general operations at 15 VA medical centers with expertise in Vascular and General surgical procedures. Assuming a recruitment rate of 3 participants per site per month, total recruitment will take approximately four years to complete. The duration of the study will be five years with four year recruitment, three months active follow up, and nine months passive follow up which will be performed by the Chairman's office in order to collect 1-year post-randomization data on all-cause mortality.

Study Population: The study will include a) patients who undergo open (non-endovascular) PAD - related operations, and b) patients who undergo selected major Vascular and General Surgery operations and have prior history of PAD or IHD. Vascular Surgery operations examined will include, but not be limited to, PAD-related: aortobifemoral or aortobiiliac bypass, open abdominal aortic aneurysm repair with simultaneous repair of aortoiliac occlusive disease, visceral bypass, iliofemoral bypass, femoral bypass or endarterectomy, infrainguinal bypass, supra-aortic trunk bypass or endarterectomy, carotid endarterectomy, and major lower extremity amputations (transfemoral, through the knee, or transtibial); Other vascular surgeries: open aneurysm repair (including but not limited to carotid, subclavian, abdominal aortic, iliac, femoral, or popliteal aneurysms); and complex endovascular aneurysm repair (defined as fenestrated endograft, or endograft with need for iliac conduit, or endovascular aneurysm repair with simultaneous femoral artery reconstruction or bypass). General Surgery operations examined will include open cholecystectomy or other complex biliary reconstruction (such as open common bile duct exploration for stones, reconstruction as part of oncologic operations such as palliative pancreatic cancer procedures) , small bowel resection, pancreatectomy, colon resection, rectal resection, splenectomy, transhiatal esophagectomy, liver resection, and open ventral hernia repair. Patients will be included in the study if their postoperative Hb falls below 10gm/dl within 15 days after surgery. Intervention: Liberal transfusion strategy is the conventional transfusion method for the surgical procedures the investigators will include in the study, and is defined as transfusion when the postoperative Hb drops below 10gm/dl, with a goal to maintain Hb above 10 gm/dl. Restrictive transfusion strategy will be defined as transfusion when the postoperative Hb drops below 7gm/dl with goal to maintain Hb above 7 gm/dl.

Significance: The proposed CSP# 599 study is uniquely positioned to address the knowledge gap of postoperative transfusion thresholds in high cardiac risk patients undergoing major surgical interventions, who are currently transfused based on data from patient populations with different risk profile. The study will include patients with high IHD burden, a population that should be the most likely to benefit from a liberal transfusion strategy and CSP#599 will examine this hypothesis directly. Conversely, if the proposed trial demonstrates that this high cardiac risk patient population can tolerate restrictive transfusion well, then the results will be easy to generalize to other patient populations and the question of transfusion thresholds will be definitively addressed. Thus, the investigators believe that regardless of outcome this trial will have significant clinical and policy implications, and will substantially impact the VA and national transfusion-related guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Males and females older than 18 years of age who have postoperative Hb < 10gm/dl within 15 days after the index operation
* Patients who undergo an operation in either one of the three following categories:

  * Veterans who undergo PAD - related operations including but not limited to the following:

    * aortobifemoral or aortobiiliac bypass
    * open abdominal aortic aneurysm repair with simultaneous repair of aortoiliac occlusive disease
    * visceral bypass
    * iliofemoral bypass
    * femoral bypass or endarterectomy
    * infrainguinal bypass
    * thromboembolectomy
    * supra-aortic trunk bypass or endarterectomy
    * carotid endarterectomy
    * major lower extremity amputations (transfemoral, through the knee, or transtibial)
  * Veterans with past medical history of ischemic stroke or IHD or PAD who undergo the following general surgery procedures, defined as:

    * known prior MI
    * ECG findings consistent with prior MI
    * prior percutaneous coronary intervention
    * prior coronary artery bypass surgery
    * history of angina for which the patient is currently receiving treatment
    * stress test indicating myocardial ischemia
    * who undergo the following General Surgery operations:

      * Open cholecystectomy or other complex biliary reconstruction
      * such as open common bile duct exploration for stones
      * reconstruction as part of oncologic operations such as palliative pancreatic cancer procedures)
    * small bowel resection
    * pancreatectomy
    * colon resection
    * rectal resection
    * splenectomy
    * transhiatal esophagectomy
    * liver resection
    * gastric resection
    * open ventral hernia repair
    * Colostomies (reversals and takedowns)
    * Intestinal anastomosis takedowns and revisions
    * Gastric bypass
    * Adrenalectomies
    * Major diaphragmatic hiatal hernia repairs
  * Veterans with past medical history of ischemic stroke or IHD or PAD who undergo the following Vascular Surgery operations:

    * Open aneurysm repair, including but not limited to:

      * carotid
      * subclavian
      * abdominal aortic
      * iliac
      * femoral
      * popliteal aneurysms
    * and complex endovascular aneurysm repair, defined as:

      * fenestrated endograft
      * or endograft with need for iliac conduit
      * or endovascular aneurysm repair with simultaneous femoral artery reconstruction or bypass
    * Subclavian/vertebral bypasses and transpositions
* Patients undergoing the above procedures will be included in the study regardless of their preoperative Hb level, and regardless of preoperative or intraoperative transfusion they might have received.

Exclusion Criteria:

* Veteran unable to consent
* Veteran unwilling to follow protocol (such as Jehovah's witnesses)
* Veteran with known history of hereditary anemias such as Thalassemia or Sickle cell disease
* Veteran with known history of hereditary bleeding disorders, such as factor VIII or factor IX deficiency
* Veteran with prior history of adverse reaction to blood administration, such as fever, rash, or hemolysis
* Veteran does not speak or understand English
* Veteran hemodynamically unstable or in cardiogenic shock for >48 hours after the index procedure
* Veteran participating in another interventional trial whose objective is to evaluate the effect of transfusion on outcomes
* Pregnancy in female Veterans
* Veteran is a prisoner or in custody of law enforcement
* Prior randomization in the CSP#599
* Patients who are known to have tested positive for COVID-19 and have not recovered prior to consent will not be consented. Any participant who is known to have a positive COVID-19 test during the screening process and has not recovered will be excluded prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1424 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2024-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis Kougias, MD MSc, Study Chair — VA New York Harbor Health Care System, Brooklyn Campus
Locations (16):
- United States (16):
  - Central Arkansas VHS John L. McClellan Memorial Veterans Hospital, Little Rock, AR, Little Rock, Arkansas
  - VA Loma Linda Healthcare System, Loma Linda, CA, Loma Linda, California
  - VA Long Beach Healthcare System, Long Beach, CA, Long Beach, California
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California
  - North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida
  - James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - VA Western New York Healthcare System, Buffalo, NY, Buffalo, New York
  - Asheville VA Medical Center, Asheville, NC, Asheville, North Carolina
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kougias P, Sharath SE, Zhan M, Carson JL, Norman LE, Mi Z, Pal R, Dosluoglu H, Modrall JG, Sarosi GA Jr, Nelson P, Arya S, Scrymgeour A, Ollison J, Calais LA, Nambi V, Gregg LP, Abdullah SM, Tsai S, Becker N, Choi JC, Chiu L, Scali S, Barshes NR, Awad S, Moursi M, Koopmann MC, Sally M, Ihnat D, Ramaswamy A, Gasper W, Tzeng E, Wilson MA, Tang G, Huang G, Biswas K; TOP Trial Investigators. Liberal or Restrictive Postoperative Transfusion in Patients at High Cardiac Risk: The TOP Randomized Clinical Trial. JAMA. 2025 Dec 23;334(24):2197-2207. doi: 10.1001/jama.2025.20841. PMID 41205227
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Fergusson DA, Pagano MB, Roubinian NH, Turgeon AF, Valentine S, Trivella M, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2025 Oct 20;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub6. PMID 41114449
- [Derived] Kougias P, Mi Z, Zhan M, Carson JL, Dosluoglu H, Nelson P, Sarosi GA Jr, Arya S, Norman LE, Sharath S, Scrymgeour A, Ollison J, Calais LA, Biswas K. Transfusion trigger after operations in high cardiac risk patients (TOP) trial protocol. Protocol for a multicenter randomized controlled transfusion strategy trial. Contemp Clin Trials. 2023 Mar;126:107095. doi: 10.1016/j.cct.2023.107095. Epub 2023 Jan 20. PMID 36690072
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Trivella M, Roubinian N, Fergusson DA, Triulzi D, Doree C, Hebert PC. Transfusion thresholds for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2021 Dec 21;12(12):CD002042. doi: 10.1002/14651858.CD002042.pub5. PMID 34932836

RESULTS

PARTICIPANT FLOW:
Groups:
- Restrictive: Blood transfusion trigger: Hb<7gm/dl
- Liberal: Blood transfusion trigger: Hb<10gm/dl
Period: Overall Study
Arm/Group | Restrictive | Liberal
Started | 712 | 712
Completed | 667 | 636
Not Completed | 45 | 76

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Restrictive | Liberal | Total
Number analyzed (Participants) | 712 | 712 | 1424
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.2 (7.71) | 69.7 (8.15) | 69.9 (7.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 22 | 31
  Male | 703 | 690 | 1393
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33 | 25 | 58
  Not Hispanic or Latino | 663 | 667 | 1330
  Unknown or Not Reported | 16 | 20 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 13 | 21
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 5 | 5 | 10
  Black or African American | 125 | 143 | 268
  White | 548 | 522 | 1070
  More than one race | 6 | 4 | 10
  Unknown or Not Reported | 18 | 24 | 42

OUTCOME MEASURES:

1. Primary Outcome: A Composite Endpoint of All-cause Post-randomization Mortality, Myocardial Infarction (MI), Coronary Revascularization, Acute Renal Failure, or Post-randomization Ischemic Stroke up to 90 Days After Randomization
Description: MI will be defined using the Third Universal Definition of Myocardial Infarction. Acute renal failure will be defined as Acute Kidney Injury stage III according to RIFLE criteria. Baseline creatinine will be considered the creatinine upon admission prior to the index operation. The above urine output criteria will be only used for patients who are in the ICU and have precise monitoring of their urinary output. For patients on the surgical floor only serum creatinine changes will be used for assessment of this endpoint. Coronary revascularization will be defined as a coronary artery bypass graft, or percutaneous coronary intervention (either angioplasty or stenting). Stroke will be defined as new unilateral neurological deficit that lasts for more than 24 hours, and is confirmed by a brain imaging modality (computed tomography or magnetic resonance imaging study) demonstrating new brain infarct.
Time Frame: 90 days after randomization
Population: Intent to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Restrictive | Liberal
Number analyzed (Participants) | 700 | 670
Participants | 71 | 61
Statistical Analysis 1: Comparison: Restrictive vs Liberal; Test type: Superiority; p = 0.515, Chi-squared; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.62 to 1.27] — Liberal vs. restrictive arm comparison

2. Secondary Outcome: A Composite Endpoint of Postoperative Infectious Complications at 90 Days Post-randomization: Infectious Complications Will Include Wound Infections, Pneumonia, and Sepsis
Description: Wound infection will be defined according to the Centers for Disease Control and Prevention (CDC) guidelines as a) positive wound culture, or b) drainage of pus from a wound, or c) suspicion of wound infection that was drained operatively.
  Pneumonia will be defined according to the CDC definition as chest radiograph with new or progressive infiltrate, consolidation, cavitation, or pleural effusion and any of the following: new onset of purulent sputum or change in character of sputum, or organism isolated from blood culture, trans-tracheal aspirate, bronchial brushings, or biopsy.
  Sepsis will be defined as a combination of two of the following systemic inflammatory response syndrome (SIRS) criteria, plus suspected or present source of infection. SIRS criteria will include the following: temperature greater than 38C, heart rate greater than 90 beats/min, WBC > 12,000 or < 4,000, or > 10% bands.
Time Frame: 90 days after randomization
Population: Intent to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Restrictive | Liberal
Number analyzed (Participants) | 679 | 652
Participants | 100 | 103
Statistical Analysis 1: Comparison: Restrictive vs Liberal; Test type: Superiority; p = 0.587, Chi-squared; Odds Ratio (OR) = 1.09, 99% CI 2-sided [0.73 to 1.61] — Liberal vs. Restrictive arm comparison

3. Secondary Outcome: A Composite Endpoint of Cardiac Complications (Other Than MI) at 90 Days Post-randomization: Cardiac Complications Include New Cardiac Arrhythmias That Necessitate New Treatment, New or Worsening Congestive Heart Failure, and Non Fatal Cardiac Arrest
Description: The diagnosis of cardiac arrhythmias will be based on EKG findings. Only arrhythmias that result in initiation of new treatment regimen (to include medications, implantable devices, or surgical intervention) during hospitalization will be recorded.
  CHF will require at least one of the following symptoms or signs new or worsening: dyspnea at rest, orthopnea, or paroxysmal nocturnal dyspnea and radiological evidence of heart failure or worsening heart failure and increase/initiation of established treatment.
  Cardiac arrest will be defined as the cessation of cardiac pump function activity that results in loss of consciousness and absence of circulating blood flow as evidenced by absent carotid pulse. Only episodes of cardiac arrest that are reversed will be collected under this endpoint. If they are not reversed the event will be categorized as death.
Time Frame: 90 days after randomization
Population: Intent to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Restrictive | Liberal
Number analyzed (Participants) | 678 | 647
Participants | 67 | 38
Statistical Analysis 1: Comparison: Restrictive vs Liberal; Test type: Superiority; p = 0.007, Chi-squared; Odds Ratio (OR) = 0.57, 99% CI 2-sided [0.33 to 0.98] — Liberal vs. Restrictive arm comparison

4. Secondary Outcome: All-cause Mortality at 1 Year After Randomization
Description: The investigators will determine vital status by telephoning participants after hospital discharge, by searching the electronic medical record and the Death Ascertainment File.
Time Frame: 12 months after randomization
Population: Intent to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Restrictive | Liberal
Number analyzed (Participants) | 701 | 668
Participants | 105 | 94
Statistical Analysis 1: Comparison: Restrictive vs Liberal; Test type: Superiority; p = 0.634, Chi-squared; Odds Ratio (OR) = 0.93, 99% CI 2-sided [0.63 to 1.38] — Liberal vs. Restrictive arm comparison

5. Secondary Outcome: A Composite Endpoint of All-cause Mortality, MI, Coronary Revascularization, Acute Renal Failure, or Postoperative Ischemic Stroke
Description: A composite endpoint of all-cause mortality, MI, coronary revascularization, acute renal failure, or postoperative ischemic stroke.
Time Frame: 30 days after randomization
Population: Intent to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Restrictive | Liberal
Number analyzed (Participants) | 703 | 680
Participants | 45 | 33
Statistical Analysis 1: Comparison: Restrictive vs Liberal; Test type: Superiority; p = 0.212, Chi-squared; Odds Ratio (OR) = 0.75, 99% CI 2-sided [0.41 to 1.37] — Liberal vs. Restrictive arm comparison

6. Secondary Outcome: Length of Hospital Stay
Description: Length of hospital stay.
Time Frame: At hospital discharge, up to 1 year
Population: Intent to Treat population
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Restrictive | Liberal
Number analyzed (Participants) | 709 | 695
days | 5.0 [3.0 to 8.0] | 5.0 [3.0 to 8.0]
Statistical Analysis 1: Comparison: Restrictive vs Liberal; Test type: Superiority; p = 0.786, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: All SAEs: From randomization until the participant last study active follow up contact (~90 days). All-cause mortality: From randomization up to 12 months post-randomization. Other (not including serious) adverse events: Not collected
Description: All SAEs were assessed up to the last contact during the active follow-up of the study and includes all participants who were followed for about 90 days during the study. All-cause mortality was assessed for up to 12 months after randomization. Other (i.e., those that were not serious) Adverse Events were not monitored/assessed within this study and hence the number at risk is zero for both arms.
Arm/Group | Restrictive | Liberal
All-Cause Mortality (participants affected / at risk) | 105/701 | 94/668
Serious Adverse Events (participants affected / at risk) | 386/712 | 372/712
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Restrictive (N=712) | Liberal (N=712)
Anaemia (Blood and lymphatic system disorders) | 15 (15) | 6 (6)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 2 (2)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 24 (26) | 12 (12)
Atrial flutter (Cardiac disorders) | 4 (6) | 1 (1)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 2 (2)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 3 (3) | 6 (6)
Cardiac failure congestive (Cardiac disorders) | 42 (48) | 26 (29)
Cardiogenic shock (Cardiac disorders) | 2 (3) | 0 (0)
Coronary artery disease (Cardiac disorders) | 3 (3) | 4 (4)
Hypervolaemia (Cardiac disorders) | 6 (6) | 6 (6)
Myocardial infarction (Cardiac disorders) | 34 (35) | 30 (31)
Myocardial ischaemia (Cardiac disorders) | 7 (7) | 3 (3)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (2) | 3 (3)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia paroxysmal (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 3 (3)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal wall haematoma (Gastrointestinal disorders) | 2 (2) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Barrett's oesophagus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Duodenal perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Erosive oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 17 (18) | 19 (19)
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 3 (3) | 2 (2)
Ileus (Gastrointestinal disorders) | 3 (3) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 4 (4)
Intestinal mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 3 (3)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatic mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 4 (4)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Cardiac death (General disorders) | 9 (9) | 6 (6)
Catheter site haematoma (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 3 (3)
Cyst (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 7 (7) | 4 (4)
Impaired healing (General disorders) | 1 (1) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 3 (3)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 3 (3)
Vascular stent thrombosis (General disorders) | 1 (1) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 4 (4) | 2 (2)
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 4 (4) | 2 (3)
Bronchitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 4 (4) | 5 (5)
COVID-19 pneumonia (Infections and infestations) | 3 (3) | 2 (2)
Cellulitis (Infections and infestations) | 14 (15) | 13 (14)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 2 (2)
Clostridium difficile infection (Infections and infestations) | 9 (9) | 5 (5)
Diabetic foot infection (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Epididymitis (Infections and infestations) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Fungal oesophagitis (Infections and infestations) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 9 (9) | 9 (9)
Groin infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Incision site cellulitis (Infections and infestations) | 4 (4) | 1 (1)
Infected seroma (Infections and infestations) | 0 (0) | 1 (1)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1)
Infective aneurysm (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 4 (4) | 4 (4)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 11 (12) | 12 (12)
Pelvic abscess (Infections and infestations) | 0 (0) | 1 (1)
Penile infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 19 (19) | 19 (19)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0)
Post procedural cellulitis (Infections and infestations) | 3 (3) | 4 (4)
Postoperative abscess (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 3 (3) | 2 (2)
Prosthetic valve endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Scrotal abscess (Infections and infestations) | 0 (0) | 1 (1)
Scrotal cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 25 (25) | 33 (35)
Septic pulmonary embolism (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 2 (2) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Splenic abscess (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 10 (10) | 15 (16)
Vascular device infection (Infections and infestations) | 0 (0) | 1 (1)
Vascular graft infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 76 (82) | 71 (78)
Wound infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anastomotic haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anastomotic ulcer haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cystitis radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Exposure to SARS-CoV-2 (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 4 (5) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Graft thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision site haematoma (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Incision site impaired healing (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site ulcer (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lisfranc fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Mental status changes postoperative (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Pancreatic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Peripheral arterial reocclusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Post procedural fever (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 3 (3) | 14 (14)
Post procedural oedema (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Postoperative delirium (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Postoperative wound complication (Injury, poisoning and procedural complications) | 5 (6) | 3 (3)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Rotator cuff syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 5 (5) | 6 (6)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular graft complication (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 9 (9) | 6 (6)
Vascular graft stenosis (Injury, poisoning and procedural complications) | 7 (7) | 2 (2)
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 2 (2) | 5 (5)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Wound complication (Injury, poisoning and procedural complications) | 14 (16) | 22 (22)
Wound dehiscence (Injury, poisoning and procedural complications) | 12 (12) | 11 (12)
Wound haematoma (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound necrosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Angiocardiogram (Investigations) | 0 (0) | 1 (1)
Angiogram peripheral (Investigations) | 1 (1) | 1 (1)
Ankle brachial index decreased (Investigations) | 1 (1) | 0 (0)
Anticoagulation drug level below therapeutic (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Cardiac pacemaker evaluation (Investigations) | 0 (0) | 1 (1)
Catheterisation cardiac (Investigations) | 0 (0) | 3 (3)
Colonoscopy (Investigations) | 0 (0) | 1 (1)
Electrocardiogram ST segment abnormal (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Myocardial necrosis marker increased (Investigations) | 5 (5) | 4 (4)
Oxygen consumption increased (Investigations) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 4 (4) | 6 (6)
White blood cell count increased (Investigations) | 1 (1) | 0 (0)
Calciphylaxis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 2 (2) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Brain injury (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 8 (8) | 7 (7)
Dizziness postural (Nervous system disorders) | 2 (2) | 1 (1)
Encephalopathy (Nervous system disorders) | 2 (2) | 4 (4)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 2 (2)
Myelopathy (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 3 (3) | 0 (0)
Seizure (Nervous system disorders) | 4 (6) | 0 (0)
Spinal cord ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 4 (4) | 2 (2)
Toxic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 2 (2)
Device occlusion (Product Issues) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (2) | 0 (0)
Delirium (Psychiatric disorders) | 4 (4) | 3 (3)
Mental status changes (Psychiatric disorders) | 0 (0) | 2 (3)
Suicidal ideation (Psychiatric disorders) | 3 (4) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 32 (34) | 33 (37)
Bladder outlet obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 1 (1) | 1 (1)
Glomerulonephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 4 (4)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Scrotal swelling (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 10 (11)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (4)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Ischaemic skin ulcer (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Prosthesis user (Social circumstances) | 0 (0) | 1 (1)
Social stay hospitalisation (Social circumstances) | 5 (5) | 7 (7)
Alcohol detoxification (Surgical and medical procedures) | 1 (1) | 0 (0)
Amputation (Surgical and medical procedures) | 8 (8) | 9 (9)
Aneurysm repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Anticoagulant therapy (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic aneurysm repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Arterial repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Arterial stent insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Arteriovenous fistula operation (Surgical and medical procedures) | 3 (3) | 1 (1)
Cardiac ablation (Surgical and medical procedures) | 1 (1) | 0 (0)
Cataract operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Catheter directed thrombolysis (Surgical and medical procedures) | 0 (0) | 1 (1)
Coronary artery bypass (Surgical and medical procedures) | 3 (3) | 2 (2)
Coronary revascularisation (Surgical and medical procedures) | 3 (3) | 1 (1)
Debridement (Surgical and medical procedures) | 3 (3) | 4 (4)
Fasciotomy (Surgical and medical procedures) | 2 (2) | 0 (0)
Foot amputation (Surgical and medical procedures) | 5 (5) | 5 (5)
Gastrointestinal tube insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Gastrostomy (Surgical and medical procedures) | 1 (1) | 1 (1)
Hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Hospitalisation (Surgical and medical procedures) | 0 (0) | 1 (1)
Implantable defibrillator insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Jejunostomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Leg amputation (Surgical and medical procedures) | 17 (18) | 20 (20)
Nephrostomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Percutaneous coronary intervention (Surgical and medical procedures) | 7 (7) | 5 (5)
Peripheral artery angioplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Peripheral artery bypass (Surgical and medical procedures) | 2 (2) | 0 (0)
Peripheral revascularisation (Surgical and medical procedures) | 4 (4) | 3 (3)
Plastic surgery of the lips and mouth (Surgical and medical procedures) | 0 (0) | 1 (1)
Post procedural drainage (Surgical and medical procedures) | 1 (1) | 0 (0)
Skin graft (Surgical and medical procedures) | 1 (1) | 0 (0)
Spinal fusion surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Spinal laminectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Thrombectomy (Surgical and medical procedures) | 2 (2) | 1 (1)
Toe amputation (Surgical and medical procedures) | 9 (9) | 6 (6)
Tracheostomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Transurethral bladder resection (Surgical and medical procedures) | 1 (1) | 0 (0)
Vascular graft (Surgical and medical procedures) | 0 (0) | 1 (1)
Wound closure (Surgical and medical procedures) | 3 (3) | 3 (3)
Aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Aortic occlusion (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Atheroembolism (Vascular disorders) | 0 (0) | 1 (1)
Blue toe syndrome (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 8 (8) | 3 (3)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 2 (2)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive urgency (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 14 (14) | 3 (3)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Iliac artery occlusion (Vascular disorders) | 0 (0) | 2 (2)
Lymphocele (Vascular disorders) | 1 (1) | 1 (1)
Lymphorrhoea (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 7 (7) | 7 (7)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 3 (3)
Peripheral artery stenosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 2 (2)
Peripheral ischaemia (Vascular disorders) | 8 (8) | 7 (7)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 2 (2) | 2 (2)
Steal syndrome (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-12-18): https://cdn.clinicaltrials.gov/large-docs/41/NCT03229941/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-28): https://cdn.clinicaltrials.gov/large-docs/41/NCT03229941/SAP_001.pdf